CLINICAL TRIAL: NCT04484610
Title: Providing Appropriate Opioid Prescription Quantities for Acute Pain Treatment: A Cluster Randomized Controlled Trial.
Brief Title: Appropriate Opioid Quantities for Acute Pain - Pharmacist Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Institute of Safe Medication Practices Canada (Unknown); North York General Hospital (Other); The Royal Ottawa Mental Health Centre (Other); Ontario Drug Policy Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 002-2019
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Opioid Use; Acute Pain
Keywords: opioid; acute pain; pharmacist; pharmacy practice
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appropriate Opioid Quantities (Experimental): Pharmacists in the intervention regions are invited to complete an eLearning program to promote the practice change intervention of assessing and dispensing appropriate quantities of opioids prescribed for acute pain.
  Interventions: Drug: Pharmacist Practice Change to Dispense Appropriate Opioid Quantities for Acute Pain
- Usual Practice (No Intervention): Pharmacists in the comparison regions are not targeted for the practice change intervention (they are not invited nor provided access to the eLearning program).

INTERVENTIONS:
Drug: Pharmacist Practice Change to Dispense Appropriate Opioid Quantities for Acute Pain — Pharmacist eLearning modules, support tools and resources to promote assessing and dispensing appropriate opioid quantities for acute pain.
  Arms: Appropriate Opioid Quantities

SUMMARY:
Prescription opioids contribute to opioid related deaths, overdose and addiction. Unused prescribed opioids are not routinely being stored or disposed of appropriately and their availability is associated with harms. Maximum daily doses prescribed are higher than that recommended in a significant number of patients. This study is designed to help have appropriate doses and quantities of opioids dispensed for the treatment of short-term pain. Rather than targeting prescribing, this study targets the dispensing process by training community pharmacists to assess the appropriateness and safety of opioid prescriptions for short-term pain and to work with patients to partially fill prescriptions if the quantities prescribed are deemed excessive. Patient education tools were developed to help promote understanding of opioid safety, including the use of appropriate quantities, safe storage and safe disposal. Pharmacists in five randomly selected regions in Ontario, Canada are targeted for the eLearning intervention. The primary study outcome is the quantities dispensed for initial opioid prescriptions for short-term pain in the intervention regions compared to ten control regions.

DETAILED DESCRIPTION:
The proposed intervention is designed to implement and evaluate a pharmacist-led intervention to promote dispensing appropriate doses and quantities of opioids for acute pain at the initial prescription stage. This would include patients discharged from hospital post-surgery, following emergency room visits, after dental procedures, and patients visiting primary care prescribers. Thus it will capture a wide spectrum of prescribing. This study focuses on incorporating into routine pharmacy practice the assessment and adjustment of opioid doses and quantities for the treatment of acute pain to appropriate levels. Pharmacists in Ontario are able to reduce the quantities of prescriptions with the agreement of the patient. The remainder of the prescription quantity can remain active to be filled subsequently if needed. By implementing the option of part-fills for prescriptions with higher quantities, this intervention does allow patients to access more analgesia if their pain management requires it.

Project Objectives

1. To develop, test, optimize and implement an intervention in 5 randomly selected regions in Ontario to promote pharmacist-led practices to limit initial quantities of opioid prescriptions to appropriate levels for the treatment of acute pain. The intervention components include a pharmacist a training program, patient engagement tools and prescriber engagement communication.
2. To measure pharmacist uptake of the intervention.
3. To compare initial prescription opioid quantities and daily doses in the intervention regions to 10 matched control regions.

This is a prospective, cluster randomized controlled trial evaluating a 6-month pharmacy practice intervention to limit initial doses and quantities of opioid prescriptions to appropriate levels for the treatment of acute pain. The intervention components include a pharmacist a training program, patient engagement tools and prescriber engagement communication. The development of the intervention was informed by the systematic approach described by French and colleagues (2012) for behaviour change interventions implementing evidence into practice. The 5 eLearning modules (15-20 minutes each) and the patient communication tools (patient handout and pharmacy poster) have undergone usability testing using a human factors research approach prior to finalization. The intervention will be implemented in 5 public health unit regions in Ontario randomly selected along with 10 matched (1:2) control public health unit regions. All community pharmacists in the intervention regions will be invited to undertake the eLearning program to promote the specific practice change related to opioid quantities. The primary outcome measure will be the quantities of opioids dispensed to patients receiving initial prescriptions for the treatment of acute pain. Analyses will be at the cluster level in which quantities dispensed will be compared both between intervention and control public health unit regions after 6 months, and before and after implementation within intervention sites.

ELIGIBILITY:
Inclusion Criteria:

* Any pharmacist working in a community pharmacy in the intervention regions.
* Any patient seeking to fill an opioid prescription for acute pain at a pharmacy in the intervention regions.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Opioid Quantities Dispensed | 6 months
  Quantities dispensed for initial opioid prescriptions from all pharmacies within the 5 intervention regions for all patients without previous opioid prescriptions in the last 6 months.

SECONDARY OUTCOMES:
Opioid Doses Dispensed | After 6 months
  Percentage of patients who were newly dispensed an opioid prescription greater than 50 milligram morphine equivalents (MME) per day.
Subsequent Opioid Dispensing | 6 months
  Frequency of dispensing remaining quantities from part-filled prescriptions and ongoing opioid dispensing.
Opioid Quantity Changes per Pharmacy, Pharmacist and Prescriber | 6 months
  Number of pharmacies, pharmacists and prescribers for which there were significant pre-post intervention changes in opioid quantities.
Prescription costs | 6 months
  Prescription cost changes related to dispensing smaller quantities: exploring the potential decreases in drug costs associated with reduced quantities, as well as potential increases in prescription costs related to extra dispensing fees for part-fill prescriptions requiring subsequent fills.
Indication for opioid | 6 months
  Types of indications for opioid prescriptions.
Pharmacists opinions, attitudes, comfort level and actions | Before and after opioid quantity education and after 6 months
  Survey
Patient experiences | After interaction with pharmacist.
  Survey
Prescriber experiences | After 6 months
  Survey

CONTACTS AND LOCATIONS:
Overall Officials: Beth Sproule, PharmD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Beth Sproule, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No